CLINICAL TRIAL: NCT06490510
Title: Prognostic Significance of Mutation Type and Chromosome Fragility in Fanconi Anemia
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PFA-2024-47
Record Dates: First submitted 2024-05-17; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to analyze the data included in the Spanish Registry of Patients with Fanconi anemia to better understand the natural history of the disease, identify genetic risk and prognostic factors, and identify potential therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Spanish Registry of Patients with Fanconi Anemia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fanconi anemia included in the Spanish Registry
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Description of the clinical evolution of the patient | 1 month
  Study the clinical evolution of patients with Fanconi anemia

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Surrallés, PhD, Principal Investigator — Institut de Recerca Sant Pau (IR SANT PAU), Barcelona, Spain
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau - IIB Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Ramirez MJ, Pujol R, Minguillon J, Bogliolo M, Persico I, Cavero D, de la Cal A, Rio P, Navarro S, Casado JA, Bailador A, de la Fuente AS, de Heredia ML, Almazan F, Antelo ML, Argiles B, Badell I, Baragano M, Belendez C, Bermudez M, Bernues M, Buedo MI, Carrasco E, Catala A, Costa D, Cuesta I, Fernandez-Delgado R, Fernandez-Teijeiro A, Figuera A, Garcia M, Gondra A, Gonzalez M, Muniz SG, Hernandez-Rodriguez I, Ibanez F, Kelleher NJ, Lendinez F, Lopez M, Lopez-Almaraz R, Marchante I, Mendoza C, Nieto J, Ojeda E, Payan-Pernia S, Pelaez I, de Soto IP, Portugal R, Ramos-Arroyo MA, Regueiro A, Rodriguez A, Rosell J, Saez R, Sanchez J, Sanchez M, Senent M, Tapia M, Trujillo-Quintero JP, Vagace JM, Verdu-Amoros J, Verdugo V, Vidales I, Villarreal J, Diaz-de-Heredia C, Sevilla J, Bueren JA, Surralles J. Prognostic significance of mutation type and chromosome fragility in Fanconi anemia. Am J Hematol. 2025 Feb;100(2):272-284. doi: 10.1002/ajh.27520. Epub 2024 Nov 19. PMID 39562502